CLINICAL TRIAL: NCT01196923
Title: Post-Market Clinical Study of the CardioFocus Endoscopic Ablation System - Adaptive Contact (CF-EAS-AC) for the Treatment of Symptomatic Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-2858
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

ARMS (1):
- HeartLight Ablation (Experimental)
  Interventions: Device: Endoscopically Guided Ablation

INTERVENTIONS:
Device: Endoscopically Guided Ablation — Visually Guided Ablation using EAS-AC

SUMMARY:
The purpose of this study is to confirm the safety and effectiveness of the CardioFocus Endoscopic Ablation System with Adaptive Contact in the treatment of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, Paroxysmal Atrial Fibrillation (AF)
* 18 to 70 Years of age
* Others

Exclusion Criteria:

* Generally good overall health as determined by multiple criteria
* Willing to participate in a study
* Others

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burke Barrett, Study Director — CardioFocus
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- HeartLight Ablation: Pulmonary Vein Isolation with the HeartLight System
Period: Overall Study
Arm/Group | HeartLight Ablation
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HeartLight Ablation: Pulmonary Vein Isolation with the HeartLight System. Participants with data available are reported so that not all measures may include data from 20 participants.
Arm/Group | HeartLight Ablation
Number analyzed (Participants) | 20
Age, Customized [Mean (Full Range); unit: years]
  Average age, reported data | 59 [43 to 74]
Gender [Number; unit: participants with data available]
  Female | 3
  Male | 16
Region of Enrollment [Number; unit: participants]
  Italy | 20

OUTCOME MEASURES:

1. Primary Outcome: Acute Isolation of Pulmonary Veins.
Description: 99% of pulmonary veins were isolated (72/73)
Time Frame: Acute PVI measured on the day of treatment
Population: All treated participants with reported data.
Measure: Number; unit: percent isolated pulmonary veins
Arm/Group | HeartLight Acutely Isolated Pulmonary Veins
Number analyzed (Participants) | 20
percent isolated pulmonary veins | 99

ADVERSE EVENTS:
Time Frame: Acute, peri-procedural assessment of adverse events.
Arm/Group | HeartLight Ablation
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartLight Ablation (N=20)
Pericardial effusion (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No